CLINICAL TRIAL: NCT01431469
Title: Efficacy and Tolerance of a Follow-On Formula Fed to Children From 12-48 Months of Age in Salvador, Bahia, Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Federal University of Bahia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6001
Record Dates: First submitted 2011-08-31; First posted 2011-09-09 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Acute Respiratory Infection; Diarrheal Disease
MeSH Terms: interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Cow's Milk (Placebo Comparator): Powdered Whole Cow's Milk
  Interventions: Dietary Supplement: Cow's milk
- Follow-On Formula (Experimental): Powdered Follow-On Formula with added long-chain Polyunsaturated fatty acid, prebiotics, and polysaccharide
  Interventions: Dietary Supplement: Follow-On Formula

INTERVENTIONS:
Dietary Supplement: Cow's milk — Powdered Whole Cow's Milk
  Arms: Cow's Milk
Dietary Supplement: Follow-On Formula — Powdered Follow-On Formula with added long-chain Polyunsaturated fatty acid, prebiotics, and polysaccharide
  Arms: Follow-On Formula

SUMMARY:
The purpose is to determine if the consumption of study product has an effect on acute respiratory infections and/or diarrheal disease.

ELIGIBILITY:
Inclusion Criteria:

* Child 12-48 months of age
* Has consumed cow's milk or a cow's milk-based beverage during the 48 hours prior to randomization
* Signed informed consent

Exclusion Criteria:

* Child who is receiving predominantly breast-milk
* Child who received any food product or supplement containing probiotics or prebiotics in the 15 days prior to randomization
* Child with allergy to gluten or serious concurrent illness that will interfere in the general management of the child
* Child with diarrhea or acute respiratory infection during the 48 hours prior to randomization
* Child's z-score of weight for length/height < -3 according to World Health Organization criteria

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Episodes of acute respiratory infections and diarrheal disease | 28 weeks

SECONDARY OUTCOMES:
Occurrence of allergic manifestations | 28 weeks
Systemic antibiotic use | 28 weeks
Duration of acute respiratory infection and diarrheal disease | 28 weeks
Changes in stool patterns | 28 weeks
Fecal and serum immune markers | 28 weeks
Serum Ferritin and Zinc status | 28 weeks
Incidence of stool parasites | 28 weeks
Growth | 28 weeks
Incidence of adverse events | 28 weeks
  The incidence of any adverse event for each participant
Acceptance of study product | 28 weeks
  Acceptance of study product based on quantity consumed

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal da Bahia, Hospital Universitário Prof. Edgard Santos Complexo HUPES, Centro Pediátrico Professor Hossanah Oliveira, Centro da Pesquisas Fima Lifshitz, Rua Augusto Viana s/n Canela, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Pontes MV, Ribeiro TC, Ribeiro H, de Mattos AP, Almeida IR, Leal VM, Cabral GN, Stolz S, Zhuang W, Scalabrin DM. Cow's milk-based beverage consumption in 1- to 4-year-olds and allergic manifestations: an RCT. Nutr J. 2016 Feb 27;15:19. doi: 10.1186/s12937-016-0138-0. PMID 26920136